CLINICAL TRIAL: NCT01362192
Title: A Clinical Evaluation of the Treatment of Lower Extremity Spider Veins Using a Dual Wavelength Laser Emitting 532 nm and 1064 nm Laser Energy
Brief Title: Treatment of Lower Extremity Spider Veins With Excel V
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-11-XLV01
Record Dates: First submitted 2011-05-25; First posted 2011-05-30 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Telangiectasis; Spider Veins
Keywords: Telangiectasis; Spider Veins; Excel V; Cutera; Laser; Leg Veins; Venulectasia; Lower Extremity veins; Laser light; KTP; 532nm
MeSH Terms: conditions — Telangiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 532 nm KTP Laser Treatment (Other)
  Interventions: Device: 532 nm KTP Excel V Laser, manufactured by Cutera, Inc.

INTERVENTIONS:
Device: 532 nm KTP Excel V Laser, manufactured by Cutera, Inc. — The 532 nm KTP Excel V laser treatment parameters to be used in this study are as follows:
  * Spot Size: 5 mm
  * Fluence: 13-15 J/cm2
  * Pulse Duration: 40 ms
  * Epidermal contact-cooling: 5° Celsius
  Other Names: Excel V laser; ExcelV; KTP; 532nm

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a new laser for the removal of unsightly spider veins on the legs. The device used in this study is the Cutera Excel V laser, which is a dual wavelength 532 nm potassium titanyl phosphate (KTP) and 1064 nm neodymium-doped yttrium aluminum garnet (Nd:YAG) laser. The Excel V laser has received 510(k) clearance from the FDA, which means the FDA has approved the laser for dermatological and vascular conditions, like spider veins.

DETAILED DESCRIPTION:
Each subject will receive 532 nm KTP laser treatment for their lower extremity spider veins in at least 2, and up to 4, separate areas. Subjects will receive 2 laser treatments spaced 12 weeks apart. Subjects will be followed for 24 weeks (12 weeks after the final laser treatment). Efficacy will be evaluated by blinded independent physician assessment of improvement in treated spider veins using digital photographs taken at baseline and the final follow-up visit by a third-party medical photography service. In addition, efficacy will be evaluated by the Investigator's mean global assessment of improvement and the subject's mean assessment of improvement. Safety will be evaluated by continuous monitoring of adverse events (AEs) and measuring pain associated with laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I - III
* Having at least 2 separate areas measuring 5cm x 5cm of lower extremity spider veins
* Having lower extremity spider veins less than 2.0mm in diameter, linear or branching, and red, pink, blue and/or purple in color, as assessed by the Investigator
* Having lower extremity spider veins appropriate for laser treatment, as assessed by the Investigator
* Subject must be able to read, understand and sign the Informed Consent Form
* Subject must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions
* Wiling to have limited sun exposure for the duration of the study, including the follow-up period
* Willingness to have digital photographs taken of lower extremity spider veins
* Agree not to undergo any other procedure for the treatment of lower extremity spider veins during the study
* Willing to not take any 'prn' medications for aches and pains (such as Tylenol® or Advil®) on the days of the laser treatments
* For female candidates - post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study

Exclusion Criteria:

* Having received any prior laser treatment for lower extremity spider veins
* Fitzpatrick Skin Type IV - VI
* Pregnant
* Having an infection, dermatitis or a rash in the treatment area
* Having significant varicosities or perforator veins
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation
* Having a known anticoagulative condition or taking anticoagulation medications
* History of thromboembolic disease, such as deep vein thrombosis (DVT)
* History of seizure disorders due to light
* Having a history of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area, unless treatment is conducted following a prophylactic regimen
* Having undergone any surgery in the treatment area within 6 months of treatment (or more if skin has not healed completely)
* Suffering from significant concurrent illness, such as insulin-dependent diabetes (type I or II), peripheral vascular disease or peripheral neuropathy
* Undergoing systemic chemotherapy for the treatment of cancer
* Systemic use of isotretinoin (Accutane®) within 6 months of study participation
* Any use of gold therapy for disorders such as rheumatologic disease or lupus
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study
* Participation in a study of another device or drug within three months prior to enrollment or during the study
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Main Line Center for Laser Surgery, Ardmore, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 532 nm KTP Laser Treatment: Each subject will receive 532 nm KTP laser treatment for their lower extremity spider veins
Period: Overall Study
Arm/Group | 532 nm KTP Laser Treatment
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 48 [32 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Fitzpatrick Skin Type [Number; unit: participants] — The Fitzpatrick Skin Type is a skin classification system based on color, genetics and reaction to sun exposure. Types range from the I to VI, where type I represents very fair-skinned individuals and type VI represents very dark-skinned individuals.
  participants
    I | 1
    II | 15
    III | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Improvement of Lower Extremity Spider Veins Based on Blinded Photo Assessments
Description: A panel of independent physicians will assess before and after digital photographs of each treated area. The physicians will be blinded to the treatment parameters and to the temporal order of the before and after photographs. Each independent physician will be asked to select the baseline photograph for each treated area and then rate the degree of improvement using the following scale:
  * 0 = No Improvement (0%)
  * 1 = Mild Improvement (< 25%)
  * 2 = Moderate Improvement (26 to 50%)
  * 3 = Significant Improvement (51 to 75%)
  * 4 = Very Significant Improvement (76 to 100%)
Time Frame: 24 weeks (12 weeks post-final laser treatment)
Population: per protocol
Measure: Mean (95% Confidence Interval); unit: points on Improvement scale
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 16
points on Improvement scale | 2.5 [1.9 to 2.9]

2. Secondary Outcome: Mean Improvement of Lower Extremity Spider Veins Based on Blinded Photo Assessments
Description: The panel of independent physicians will be asked to select the baseline photograph for each treated area and then rate the degree of improvement using the following scale:
  * 0 = No Improvement (0%)
  * 1 = Mild Improvement (< 25%)
  * 2 = Moderate Improvement (26 to 50%)
  * 3 = Significant Improvement (51 to 75%)
  * 4 = Very Significant Improvement (76 to 100%)
Time Frame: 12 weeks (post-1st laser treatment)
Population: per protocol
Measure: Mean (95% Confidence Interval); unit: points on Improvement scale
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 16
points on Improvement scale | 1.8 [1.0 to 2.4]

3. Secondary Outcome: Percent of Subjects With "Significant" or "Very Significant" Improvement in Lower Extremity Spider Veins, as Assessed by the Treating Investigator.
Description: The Investigator will perform the Physician's Global Assessment of the degree of improvement for each treated area of the subject's lower extremity spider veins using the following scale:
  * 0 = No Improvement (0%)
  * 1 = Mild Improvement (< 25%)
  * 2 = Moderate Improvement (26 to 50%)
  * 3 = Significant Improvement (51 to 75%)
  * 4 = Very Significant Improvement (76 to 100%)
Time Frame: 24 weeks (12 weeks post-final laser treatment)
Population: per protocol
Measure: Number; unit: percent of participants
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 16
percent of participants | 69

4. Secondary Outcome: Percent of Subjects With "Significant" to "Very Significant" Improvement of Lower Extremity Spider Veins, as Assessed by Subject.
Description: Subjects will be asked to rate the improvement of each treated area of their lower extremity spider veins as compared to baseline using the following scale:
  * 0 = No Improvement (0%)
  * 1 = Mild Improvement (< 25%)
  * 2 = Moderate Improvement (26 to 50%)
  * 3 = Significant Improvement (51 to 75%)
  * 4 = Very Significant Improvement (76 to 100%)
Time Frame: 24 weeks (12 weeks post-final laser treatment)
Population: per protocol
Measure: Number; unit: percent of participants
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 16
percent of participants | 75

5. Secondary Outcome: Percent of Subjects Satisfied With Improvement of Treated Spider Veins.
Description: Subjects will assess their satisfaction with the procedure and with the improvement in lower extremity spider veins at twelve weeks post final laser treatment based using the following scale:
  * 1 = Very Much Not Satisfied
  * 2 = Not Satisfied
  * 3 = Somewhat Satisfied
  * 4 = Satisfied
  * 5 = Very Much Satisfied
Time Frame: 24 weeks (12 weeks post-final laser treatment)
Population: per protocol
Measure: Number; unit: percent of participants
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 16
percent of participants | 100

6. Secondary Outcome: Mean Pain Score Associated With Laser Treatment.
Description: Subjects will be asked to rate the average pain experienced during laser treatments using the 0-10 numeric pain rating scale (0 = no pain to 10 = worst possible pain).
Time Frame: Day 0 (1st laser treatment)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: Numeric Pain Rating Score
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 20
Numeric Pain Rating Score | 3.2 (1.0)

7. Secondary Outcome: Mean Pain Score Associated With Laser Treatment
Description: as for outcome 6
Time Frame: 12 weeks (2nd laser treatment)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: Numeric Pain Rating Score
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 20
Numeric Pain Rating Score | 2.5 (0.9)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | 532 nm KTP Laser Treatment
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 532 nm KTP Laser Treatment (N=20)
Post-Inflammatory Hyperpigmentation at 24 weeks (Skin and subcutaneous tissue disorders) | 1 (1)
Mild Edema Immediate Post-TX #1 (Skin and subcutaneous tissue disorders) | 7 (7)
Mild Erythema Immediate Post-TX#1 (Skin and subcutaneous tissue disorders) | 11 (11)
Moderate Erythema Post-TX#1 (Skin and subcutaneous tissue disorders) | 8 (8)
Mild Edema Immediate Post-TX#2 (Skin and subcutaneous tissue disorders) | 8 (8)
Moderate Edema Immediate Post-TX#2 (Skin and subcutaneous tissue disorders) | 1 (1)
Mild Erythema Post-TX#2 (Skin and subcutaneous tissue disorders) | 13 (13)
Moderate Erythema Post-TX#2 (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No